CLINICAL TRIAL: NCT06038825
Title: The Effect of Topical Vibration on Injection Pain in Scalp Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, derya özkan, professor medical doctor, Diskapi Teaching and Research Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: scalp block
Record Dates: First submitted 2023-08-01; First posted 2023-09-15 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Analgesia
Keywords: scalp clock; awake craniotomy; vibration
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- topical vibration (Active Comparator): For all patients one half of the scalp was injected with vibration device.
  Interventions: Device: topical vibration
- control (No Intervention): Same patient's other side of the scalp was injected without vibration device.

INTERVENTIONS:
Device: topical vibration — topical vibration (Aprilla brand, giving 6000 vibrations per minute) is a device for pain relief during injection of local anesthetic.
  Arms: topical vibration

SUMMARY:
In this study; it's aimed to reduce injection pain during the practice of scalp block, which is used as a method of anesthesia in patients who underwent awake craniotomy surgery. For this purpose, the investigators used topical vibration stimulation, which is non-invasive procedure.

DETAILED DESCRIPTION:
Scalp block is an analgesia technique frequently used in neurosurgical procedures. In this block, while providing adequate anesthesia for surgery, it also helps to preserve hemodynamics by inhibiting pain sensation. In this block, there is a certain degree of pain due to multiple injections. The transmission of pain sensation to the cortex is reduced by costimulating the receptors that transmit the pain sensation with vibration stimulus. In this study; it was aimed to investigate the effect of topical vibration on injection pain in participants who received sedoanalgesia with dexmedetomidine in bilateral scalp block practice.

In routine clinical practice, bilateral scalp block (local anesthetic injection into greater occipital, lesser occipital, supratrochlear, supraorbital, auriculotemporal, zygomaticotemporal nerves) is performed in participants who is sedated. While local anesthetic is injecting, vibration device (Aprilla brand, giving 6000 vibrations per minute) will be vibrated for 10 seconds and then local anesthetic will be injected. Meanwhile, participants' numerical pain scores (NRS) and hemodynamic parameters will be monitored.

In this study, the NRS scores and hemodynamic variables of the participants will be compared during the local anesthetic application of each 6 nerves bilaterally and during the injections of the nerves with and without the use of vibration.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-75
* ASA (American Society of Anesthesiologists) Scoring I-III
* Cases in which scalp block will be applied

Exclusion Criteria:

* ASA score IV

  * Uncooperative
  * Known allergy to any of the study drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
pain score (NRS) | during needling (injection) procedure
  0 ; no pain,10; the worst pain ever possible

SECONDARY OUTCOMES:
Mean arterial pressure (mmHg) | baseline, during needling procedure, 1 min after needling
Heart Rate (beat/min) | baseline, during needling procedure, 1 min after needling

CONTACTS AND LOCATIONS:
Overall Officials: nur yilmaz, specialist, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuwahara H, Ogawa R. Using a Vibration Device to Ease Pain During Facial Needling and Injection. Eplasty. 2016 Feb 4;16:e9. eCollection 2016. PMID 26933468
- [Derived] Yilmaz N, Caparlar CO, Kilincarslan A, Sipahioglu FO, Ozkan D, Unluer C. Effect of topical vibration on pain during scalp block injections in awake craniotomy and deep brain stimulation surgery : Analgesic effects of vibratory stimulation during scalp blocks. Anaesthesiologie. 2026 Jan;75(1):20-27. doi: 10.1007/s00101-025-01604-8. Epub 2025 Nov 7. PMID 41203985